CLINICAL TRIAL: NCT01137240
Title: Assessment and Prevalence of Gastrointestinal Dysfunction in Children With Mitochondrial Disorders (MD)
Brief Title: Gastrointestinal Dysfunction in Children Affected With Mitochondrial Disorders
Status: Completed | Type: Observational
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Mary Kay Koenig, Assistant Professor - Pediatrics, The University of Texas Health Science Center, Houston
Other Study IDs: HSC-MS-10-0016
Record Dates: First submitted 2010-06-02; First posted 2010-06-04 (Estimated); Last update posted 2012-02-27 (Estimated); Status verified 2012-02

CONDITIONS: Gastrointestinal Dysfunction; Mitochondrial Disorders
Keywords: subjects suffering from mitochondrial disorders with one or more gastrointestinal symptoms would be the focus of the study
MeSH Terms: conditions — Mitochondrial Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Children with mitochondrial disorders: suffering from gastrointestinal dysfunction
  Interventions: Procedure: gastric emptying scan

INTERVENTIONS:
Procedure: gastric emptying scan — subjects will eat a solid meal (scrambled eggs, etc) or drink liquid (water or juice) mixed with approximately 0.5 millicuries of radioactive material. A scanner/external gamma camera will be placed over the subject's stomach at 15 minute intervals for a duration of 90 minutes (monitoring the amount of radioactivity in the stomach). As the radioactively-labeled food empties from the stomach, the amount of radioactivity in the stomach decreases. The rate at which the radioactivity leaves the stomach reflects the rate at which food is emptying from the stomach. The radioisotope has a half life of approximately. 6 hours and is totally eliminated from the body within 24 hours.
  In subjects with gastroparesis, the food and the attached radioactive material remain in the stomach longer than normal (usually hours) before emptying into the small intestine. As a result, the scanner continues to show radioactivity in the area of the stomach for hours after the test meal.

SUMMARY:
Hypothesis: Many patients with underlying mitochondrial disorders have feeding problems because of poor gastrointestinal motility; feeding problems lead to growth impairment and many affected children are malnourished.

DETAILED DESCRIPTION:
Specific AIM: To study gastric emptying times in children with mitochondrial disorders.

INTRODUCTION: Mitochondrial disorders are a recently described group of metabolic disorders with complex presentations; children present with a myriad of symptoms and involvement of a wide array of organ systems. Mitochondrial disorders result from dysfunction of proteins or ribosomes utilized by mitochondria. Mitochondrial dysfunction causes a lack of ATP production and without enough ATP cells are unable to perform their biological functions.

The first mitochondrial disease was described in 1962. Over the last 40 years, mitochondrial disease has become increasingly recognized as an important group of genetic disorders. The prevalence has been reported to be as high as one in 3000 children, approaching that of childhood cancer. Mitochondrial disorders have classically been described as affecting tissues with the highest demand for ATP, i.e., brain, muscles, nerves, heart, and liver. Increasing diagnosis of patients with mitochondrial disease has led to expansion of the known spectrum of systemic involvement. Many children with mitochondrial disorders have gastrointestinal manifestations, predominately constipation and poor gastrointestinal motility. Poor motility effects feeding and many of these patients are intolerant to oral feeding and require mechanical feeding to survive.

Currently there are no proven treatment strategies for children with mitochondrial disorders. Most of the current management strategies are nonspecific and target symptom control with only limited utility and success.

Study Methods: We plan to conduct a large, prospective cohort study of 25 children with mitochondrial disorders. Subjects will include children with different subclasses of various mitochondrial disease subgroups who meet the modified Walker criteria for diagnosis of a probable or definite mitochondrial disorder.

Gastric emptying times will be measured to assess gastrointestinal motility, function, and dynamics.

Research Design and Methods: Participants for this study will be recruited prospectively through the University of Texas (UT) Mitochondrial Clinic. All mitochondrial patients with probable or definite mitochondrial disorders from 3 to 18 years of age seen at the University of Texas Mitochondrial Clinic will be invited to participate. The decision to participate or not to participate in this research study will in no way affect medical care offered by clinicians involved in the UT Mitochondrial Clinic.

Consent for study participation will be obtained by the Principal Investigator (PI) or co-investigator (CI) or designated clinical nurse in person and a copy of the signed consent form will be retained on file by the PI, placed in the patient's research medical record (separate from the clinic record). For minor participation (12 to 17 years) parental permission and consent of the child will be obtained. For minor participation (7 to 11 years) parental permission and assent of the child will be obtained. For minor participation (birth to 6 years), parental permission will be obtained

This study population consists of a cohort of patients with different subsets of mitochondrial disorders, including children with isolated deficiencies of the electron transport chain and children with syndromic mitochondrial disorders. Final analysis will will evaluate results both individually and in subclass groups, ie, Complex I deficiency, MELAS (mitochondrial encephalopathy lactic acidosis and stroke-like syndrome), etc.

Research design: Patients will undergo testing for gastric emptying scans at our radiology department. The studies would be performed using Technetium-99 as tracer by our UT radiologist David Wan, MD. Patient would report on the morning of the study NPO and would drink the tracer. The transit of the contrast material through the stomach would be monitored and evaluated with regularly scheduled X Rays of the stomach and the final results would be interpreted as normal, delayed or significantly delayed.

Risks and Benefits : The risks of this study are largely confined to maintaining patient confidentiality. There will be no personal benefit to the participant/family. No payment will be offered in exchange for study participation. Successful development of a patient database will provide valuable information on the natural history of these complicated disorders.

Information derived from the database will be published in a peer reviewed medical journal; however no individual would be identified and all personal information would be kept confidential. A potential benefit to the scientific community will be greater understanding of the clinical course and expected laboratory values observed in persons with mitochondrial disease. There are no foreseeable risks to the research staff.

Confidentiality: All participants' names and other information will be kept strictly confidential. All participants will be assigned a subject ID number and an individual identification number. The code linking name and subject ID number will be maintained in a locked file in the office of the PI and in a spread sheet file on the office computer of the PI. All subsequent reference to patient data will be in anonymous form by patient identification number.

Determine if gastric emptying times in children with mitochondrial disorders are abnormal.

There are no known risks of performing gastric emptying scan studies in children.

The risk of allergy to eggs/food is similar to that observed in other children of similar age groups and is minimal.

RISKS:

Risk associated with the allergic reaction to the dye is also similar to the one observed in other children of similar age groups and is minimal.

Risk associated with breach of confidentiality- minimal. The names and other identification information pertinent to the patient's identity and test results would be strictly kept confidential and patients would be never identified by their names or other pieces of information in public or to anyone else not related to the study.

Patient's test results would also be not released to the insuring companies directly or indirectly.

Risk associated with the procedure- The procedure itself is very safe and has been performed in children of all age groups including the ones suffering from chronic disorders like the mitochondrial disorders all the time. Our radiologists are familiar with the nature of medical disorder that these children presents with and are very comfortable performing this procedure in a safe and timely manner.

ELIGIBILITY:
Inclusion Criteria:

1. Parents/Guardians are informed and given written consent.
2. Subject is willing and able to comply with all trial requirements
3. Subject is over 3 years of age.
4. Subject has a diagnosis of mitochondrial disorder validated by the modified Walker criteria used for diagnosis of mitochondrial diseases(9).
5. A female subject in the age group of 11 yrs. or older is not pregnant as evidenced by a negative urine dipstick pregnancy test
6. Subject to be enrolled has one or more of the following gastrointestinal signs and symptoms pertaining to gastrointestinal dysfunction like but not limited to abdominal pain, nausea, vomiting, bloating, indigestion, abdominal distention or sense of abdominal fullness.

Exclusion Criteria:

1. Subject is currently having one or more gastrointestinal disease/disorder that is not explained by the current knowledge of mitochondrial diseases. For example, patients suffering from peptic ulcer disease or inflammatory bowel diseases will be excluded.
2. Subject is a pregnant or a nursing female.

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: children suffering form mitochondrial disorders.
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2010-06; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jatinder Bhardwaj, MD, Principal Investigator — Privat Practice - Toledo, OH; Mary K Koenig, MD, Principal Investigator — The University of Texas Medical School at Houston
Locations (1):
- University of Texas- Houston Health Sceince Center, Houston, Texas, United States

REFERENCES:
- [Background] Koenig MK. Presentation and diagnosis of mitochondrial disorders in children. Pediatr Neurol. 2008 May;38(5):305-13. doi: 10.1016/j.pediatrneurol.2007.12.001. PMID 18410845
- [Background] Gillis LA, Sokol RJ. Gastrointestinal manifestations of mitochondrial disease. Gastroenterol Clin North Am. 2003 Sep;32(3):789-817, v. doi: 10.1016/s0889-8553(03)00052-9. PMID 14562575
- [Background] Nissenkorn A, Zeharia A, Lev D, Fatal-Valevski A, Barash V, Gutman A, Harel S, Lerman-Sagie T. Multiple presentation of mitochondrial disorders. Arch Dis Child. 1999 Sep;81(3):209-14. doi: 10.1136/adc.81.3.209. PMID 10451392